CLINICAL TRIAL: NCT03051867
Title: Vitamin D Status and Metabolism in Pregnant and Nonpregnant Control Women Consuming Controlled and Equivalent Intakes of Vitamin D
Brief Title: Vitamin D Status and Metabolism in Human Pregnancy
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: OSP 74161
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cord blood, placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Third-trimester pregnant women: Women differing in their reproductive state (pregnant versus nonpregnant) will consume equivalent dietary intakes of vitamin D and related nutrients as part of a feeding study.
- Nonpregnant control women: Women differing in their reproductive state (pregnant versus nonpregnant) will consume equivalent dietary intakes of vitamin D and related nutrients as part of a feeding study.

SUMMARY:
The purpose of the present study is to understand the effect of pregnancy on vitamin D metabolism and requirements as well as the modulatory role of the placenta in vitamin D metabolism during pregnancy. In addition, a human placental cell culture model will be employed to examine vitamin D metabolic flux in human trophoblast cells. The impact of maternal vitamin D status on maternal and fetal bone health during gestation will also be examined.

DETAILED DESCRIPTION:
Rationale

Despite mounting evidence that maternal vitamin D status is linked to pregnancy outcomes [1,2], the impact of pregnancy on vitamin D metabolism and requirement has yet to be clearly defined. In addition, although the placenta is known to express all components of the vitamin D metabolic pathway [3,4], very little is known about placental vitamin D metabolism. Moreover, although vitamin D is known to affect bone health in the nonpregnant state, the effect of maternal vitamin D status on maternal and fetal bone health in human pregnancy is unclear [5-7]. Therefore, the present study seeks to advance current understanding of vitamin D metabolism and requirements during pregnancy.

Objective and Research Questions

This study aims to examine: 1) the effect of pregnancy on a comprehensive panel of blood biomarkers of vitamin D status and metabolism; 2) the role of the placenta in modulating circulating vitamin D metabolites; and 3) the impact of maternal vitamin D status on maternal and fetal markers of bone metabolism.

Study Population, Design, and Exposure

As a secondary analysis, this study uses biological samples obtained from pregnant and nonpregnant control women who participated in a 12-wk randomized controlled trial in 2009-2010 which featured two doses of choline (i.e., 480 or 930 mg choline/d) (NCT01127022) [8]. Throughout the controlled feeding period, 26 third-trimester pregnant women and 21 nonpregnant women (both reproductive groups aged > 21 y) in a good health status consumed equivalent intakes of vitamin D (511 IU/d), calcium (1.6 g/d) and phosphorus (1.9 g/d) from the study diet and prenatal multivitamin supplement (Pregnancy Plus; Fairhaven Health LLC) for ≥ 10 weeks.

Dependent variables:

1. Blood biomarkers of vitamin D metabolism at week 0 (study-baseline) and week 10 (representing study-end)
2. Placental biomarkers of vitamin D metabolism at delivery
3. Markers of bone metabolism in maternal and fetal cord blood as well as maternal urine

Ethical considerations

The study protocol of the original RCT was approved by the Institutional Review Board for Human Study Participant Use at Cornell University and the Cayuga Medical Center where pregnant women delivered their babies. Informed consent was obtained from all participants before study entry, and the original study was registered at clinicaltrials.gov as NCT01127022. For this secondary analysis, deidentified data will be used.

Dissemination Findings

Findings from the present study will be reported in manuscripts that will be submitted for publication to a leading medical/nutrition journal in an appropriate field (i.e. nutrition, bone, placenta, and reproductive physiology). In addition, findings will be presented as abstracts, posters, and presentations at research conferences.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21-40 y
* Healthiness as assessed by health-related questionnaire, a blood chemistry profile, and a complete blood count
* Normal liver and kidney function
* Willingness to comply with the study protocol
* Singleton pregnancy (pregnant women only)

Exclusion Criteria:

* Use of tobacco, drug, or alcohol
* Use of prescription medications known to affect liver function
* Pregnancy associated complications

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of all healthy third-trimester pregnant (n=26) and nonpregnant (n=21) women who participated in the original RCT study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-01-15 (Actual); Primary Completion 2010-12-18 (Actual); Study Completion 2011-12-18 (Actual)

PRIMARY OUTCOMES:
Maternal circulating concentrations of 25-hydroxyvitamin D | Baseline (week 0; 26-29 wk gestation) and study-end (week 10; 36-39 wk gestation)
  Serum 25-hydroxyvitamin D [25(OH)D] will be measured using an isotope dilution LC-MS/MS methodology, and the effect of reproductive state on serum 25(OH)D will be examined using a linear mixed model which considers confounding factors.
Maternal circulating concentrations of 1,25-dihydroxyvitamin D | Baseline (week 0; 26-29 wk gestation) and study-end (week 10; 36-39 wk gestation)
  Plasma 1,25-dihydroxyvitamin D [1,25(OH)2D] will be measured using an EIA kit, and the effect of reproductive state on circulating 1,25(OH)2D will be examined using a linear mixed model which considers confounding factors.
Maternal circulating concentrations 24,25-dihydroxyvitamin D | Baseline (week 0; 26-29 wk gestation) and study-end (week 10; 36-39 wk gestation)
  Plasma 24,25-dihydroxyvitamin D [24,25(OH)2D] will be measured using an isotope dilution LC-MS/MS methodology, and the effect of reproductive state on circulating 24,25(OH)2D will be examined using a linear mixed model which considers potential confounders.
Placental mRNA abundance of 25-hydroxylase | Delivery
  Placental mRNA abundance of 25-hydroxylase [CYP2R1] will be measured using a qPCR, and the associations of placental CYP2R1 mRNA abundance with serum 25(OH)D will be examined using a linear mixed model which considers potential confounders.
Placental mRNA abundance of 24-hydroxylase | Delivery
  Placental mRNA abundance of 24-hydroxylase [CYP24A1] will be measured using a qPCR, and the associations of placental CYP24A1 mRNA abundance with circulating 24,25(OH)2D will be examined using a linear mixed model which considers potential confounders.
Placental 25-hydroxyvitamin D | Delivery
  25(OH)D will be measured from placental tissue using an isotope dilution LC-MS/MS methodology, and the associations of placental 25(OH)D with serum 25(OH)D as well as placental CYP2R1 mRNA abundance will be examined using a Pearson correlation test and a linear mixed model which considers potential confounders.
Placental 24,25-dihydroxyvitamin D | Delivery
  24,25(OH)2D will be measured from placental tissue using an isotope dilution LC-MS/MS methodology, and the associations of placental 24,25(OH)2D with circulating 25(OH)D and 24,25(OH)2D as well as placental CYP24A1 mRNA abundance will be examined using a Pearson correlation test and a linear mixed model which adjusts for potential confounders.

SECONDARY OUTCOMES:
Maternal circulating intact parathyroid hormone | Baseline (week 0; 26-29 wk gestation) and study-end (week 10; 36-39 wk gestation)
  Plasma intact parathyroid hormone [iPTH] will be measured using an automated immunoassay, and the relationship of maternal serum 25(OH)D with maternal iPTH will be assessed using a linear mixed model which considers potential confounders.
Maternal circulating carboxy-terminal cross-linking telopeptide of type 1 collagen | Baseline (week 0; 26-29 wk gestation), study-end (week 10; 36-39 wk gestation), and delivery
  Plasma carboxy-terminal cross-linking telopeptide of type 1 collagen [CTx] will be measured using an ELISA kit, and the relationships of maternal serum 25(OH)D with maternal CTx will be assessed using a linear mixed model which considers potential confounders.
Maternal urinary deoxypyridinoline/creatinine | Baseline (week 0; 26-29 wk gestation), study-end (week 10; 36-39 wk gestation)
  Urinary deoxypyridinoline/creatinine [DPD/Cr] will be measured using an ELISA kit, and the relationships of maternal serum 25(OH)D with maternal DPD/Cr will be assessed using a linear mixed model which considers potential confounders.
Maternal circulating osteocalcin | Baseline (week 0; 26-29 wk gestation), study-end (week 10; 36-39 wk gestation), and delivery
  Plasma osteocalcin [OC] will be measured using an ELISA kit, and the relationships of maternal serum 25(OH)D with maternal OC will be assessed using a linear mixed model which considers potential confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caudill, PhD, Principal Investigator — Cornell University
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner CL, Taylor SN, Johnson DD, Hollis BW. The role of vitamin D in pregnancy and lactation: emerging concepts. Womens Health (Lond). 2012 May;8(3):323-40. doi: 10.2217/whe.12.17. PMID 22554179
- [Background] Aghajafari F, Nagulesapillai T, Ronksley PE, Tough SC, O'Beirne M, Rabi DM. Association between maternal serum 25-hydroxyvitamin D level and pregnancy and neonatal outcomes: systematic review and meta-analysis of observational studies. BMJ. 2013 Mar 26;346:f1169. doi: 10.1136/bmj.f1169. PMID 23533188
- [Background] Ma R, Gu Y, Zhao S, Sun J, Groome LJ, Wang Y. Expressions of vitamin D metabolic components VDBP, CYP2R1, CYP27B1, CYP24A1, and VDR in placentas from normal and preeclamptic pregnancies. Am J Physiol Endocrinol Metab. 2012 Oct 1;303(7):E928-35. doi: 10.1152/ajpendo.00279.2012. Epub 2012 Aug 7. PMID 22871339
- [Background] Liu NQ, Hewison M. Vitamin D, the placenta and pregnancy. Arch Biochem Biophys. 2012 Jul 1;523(1):37-47. doi: 10.1016/j.abb.2011.11.018. Epub 2011 Dec 2. PMID 22155151
- [Background] Olausson H, Goldberg GR, Laskey MA, Schoenmakers I, Jarjou LM, Prentice A. Calcium economy in human pregnancy and lactation. Nutr Res Rev. 2012 Jun;25(1):40-67. doi: 10.1017/S0954422411000187. PMID 22894942
- [Background] Kalra P, Das V, Agarwal A, Kumar M, Ramesh V, Bhatia E, Gupta S, Singh S, Saxena P, Bhatia V. Effect of vitamin D supplementation during pregnancy on neonatal mineral homeostasis and anthropometry of the newborn and infant. Br J Nutr. 2012 Sep 28;108(6):1052-8. doi: 10.1017/S0007114511006246. Epub 2012 Jan 3. PMID 22212646
- [Background] Hashemipour S, Lalooha F, Zahir Mirdamadi S, Ziaee A, Dabaghi Ghaleh T. Effect of vitamin D administration in vitamin D-deficient pregnant women on maternal and neonatal serum calcium and vitamin D concentrations: a randomised clinical trial. Br J Nutr. 2013 Nov 14;110(9):1611-6. doi: 10.1017/S0007114513001244. Epub 2013 Apr 29. PMID 23628132
- [Background] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen F, Stabler SP, Allen RH, Caudill MA. Maternal choline intake modulates maternal and fetal biomarkers of choline metabolism in humans. Am J Clin Nutr. 2012 May;95(5):1060-71. doi: 10.3945/ajcn.111.022772. Epub 2012 Mar 14. PMID 22418088
- [Derived] Park H, Wood MR, Malysheva OV, Jones S, Mehta S, Brannon PM, Caudill MA. Placental vitamin D metabolism and its associations with circulating vitamin D metabolites in pregnant women. Am J Clin Nutr. 2017 Dec;106(6):1439-1448. doi: 10.3945/ajcn.117.153429. Epub 2017 Oct 11. PMID 29021285